CLINICAL TRIAL: NCT05421650
Title: Therapeutic Effect of Surgical Debulking of Metastatic Lymph Nodes in Cervical Cancer Stage IIICr: A Phase III, Randomized Controlled Clinical Trial
Brief Title: Therapeutic Effect of Surgical Debulking of Metastatic Lymph Nodes in Cervical Cancer Stage IIICr
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Ju-Won Roh, Principal Investigator, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGOG1047_DEBULK
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer IIICr; Bulky or multiple lymph nodes; Surgical debulking of lymph nodes; Concurrent chemoradiation therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Concurrent chemoradiation therapy (CCRT)
  Interventions: Other: CCRT
- Experimental group (Experimental): Surgical debulking of bulky or multiple lymph node + CCRT
  Interventions: Procedure: Surgical debulking of lymph nodes + CCRT

INTERVENTIONS:
Other: CCRT — CCRT
  Arms: Control group
Procedure: Surgical debulking of lymph nodes + CCRT — Surgical debulking of lymph nodes + CCRT
  Arms: Experimental group

SUMMARY:
This study is a prospective, multicenter and randomized clinical trial (DEBULK trial) to determine the therapeutic effect of surgical debulking of bulky or multiple lymph nodes before concurrent chemoradiation therapy (CCRT) in cervical cancer stage IIICr.

DETAILED DESCRIPTION:
Bulky or multiple lymph nodes metastasis in cervical cancer shows poor prognosis and can also diminish the effect of radiotherapy or concurrent chemoradiation therapy (CCRT). However, it is difficult to increase the dose of radiation and chemotherapy considering their side effects. Therefore, the objective of this study is to determine the therapeutic effect of surgical debulking of bulky or multiple lymph nodes before concurrent chemoradiation therapy (CCRT) compared to CCRT only, in cervical cancer stage IIICr. This study is a phase III, multicenter and randomized clinical trial (DEBULK trial).

* Concurrent chemoradiation therapy (CCRT)
* Surgical debulking of bulky or multiple lymph node followed by CCRT

ELIGIBILITY:
1) Inclusion Criteria

(1) Women aged ≥ 20 years and ≤ 70 years (2) Patients newly diagnosed with squamous cell carcinoma (SCC), adenocarcinoma, or adenosquamous carcinoma (3) Patients with a short-axis diameter of the pelvic LN or para-aortic LN under the renal vein of ≥ 1.5 cm or ≥ 2 LNs with a short-axis diameter ≥ 1 cm in CT or MRI (PET-CT can be used as an auxiliary tool) (4) Patients with CCRT planned as a treatment for cervical cancer (5) Patients whose competency is Eastern Cooperative Oncology Group performance score 0-1 (6) Patients who have signed the approved informed consent form for study participants (7) Patients in whom surgical debulking for LN metastasis was possible, as confirmed by radiological examination.

2) Exclusion Criteria

(1) Patients who have been diagnosed with cancer of any organ other than thyroid cancer (excluding stage 0 cancer) within the previous 5 years (2) Patients who are pregnant or plans to conceive during the clinical study period (3) Patients with any active infectious disease or incurable severe inflammation (4) Patients who cannot undergo surgery due to internal or surgical disease (5) Patients who cannot receive chemotherapy due to internal or surgical disease (6) Patients with a history of pelvic RT (7) Patients with a history of subtotal hysterectomy (8) Patients with remote metastasis other than a pelvic or para-aortic LN (e.g., lung, subclavian, and inguinal LNs)

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression-free survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall survival
Treatment-related complications | 3 years
  Treatment-related complications
False positive rate & positive predictive value of bulky or multiple LN imaging | 6 months
  To determine the accuracy of LN metastasis in imaging study

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Won Roh, Principal Investigator — CHA University Ilsan Medical Center
Locations (26):
- Aster CMI Hospital, Bengaluru, India
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
- First Obstetrics and Gynecology Clinic, "G. E. Palade" University of Medicine, Pharmacy, Science and Technology, Târgu Mureş, Romania
- South Korea (22):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Dongguk University Medical Center, Goyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangbuk-do
  - Samsung Changwon Medical Center, Changwon, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Dongnam Institute of Radiological & Medical Sciences, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul ST. Mary's Hospital, Seoul
- Ho Chi Minh City Oncology Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Jung KW, Won YJ, Kong HJ, Lee ES. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2016. Cancer Res Treat. 2019 Apr;51(2):417-430. doi: 10.4143/crt.2019.138. Epub 2019 Mar 18. PMID 30913865
- [Background] Bhatla N, Berek JS, Cuello Fredes M, Denny LA, Grenman S, Karunaratne K, Kehoe ST, Konishi I, Olawaiye AB, Prat J, Sankaranarayanan R, Brierley J, Mutch D, Querleu D, Cibula D, Quinn M, Botha H, Sigurd L, Rice L, Ryu HS, Ngan H, Maenpaa J, Andrijono A, Purwoto G, Maheshwari A, Bafna UD, Plante M, Natarajan J. Revised FIGO staging for carcinoma of the cervix uteri. Int J Gynaecol Obstet. 2019 Apr;145(1):129-135. doi: 10.1002/ijgo.12749. Epub 2019 Jan 17. PMID 30656645
- [Background] Suprasert P, Srisomboon J, Charoenkwan K, Siriaungul S, Khunamornpong S, Siriaree S, Phongnarisorn C, Lorvidhaya V. Outcomes of abandoned radical hysterectomy in patients with stages IB-IIA cervical cancer found to have positive nodes during the operation. Int J Gynecol Cancer. 2005 May-Jun;15(3):498-502. doi: 10.1111/j.1525-1438.2005.15315.x. PMID 15882176
- [Background] Abu-Rustum NR, Yashar CM, Bean S, Bradley K, Campos SM, Chon HS, Chu C, Cohn D, Crispens MA, Damast S, Fisher CM, Frederick P, Gaffney DK, Giuntoli R, Han E, Huh WK, Lurain Iii JR, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Sisodia R, Tillmanns T, Ueda S, Urban R, Wyse E, McMillian NR, Motter AD. NCCN Guidelines Insights: Cervical Cancer, Version 1.2020. J Natl Compr Canc Netw. 2020 Jun;18(6):660-666. doi: 10.6004/jnccn.2020.0027. PMID 32502976
- [Background] Song S, Kim JY, Kim YJ, Yoo HJ, Kim SH, Kim SK, Lim MC, Kang S, Seo SS, Park SY. The size of the metastatic lymph node is an independent prognostic factor for the patients with cervical cancer treated by definitive radiotherapy. Radiother Oncol. 2013 Jul;108(1):168-73. doi: 10.1016/j.radonc.2013.04.015. Epub 2013 May 14. PMID 23684584
- [Background] Oh J, Seol KH, Choi YS, Lee JW, Bae JY. Clinical significance of lymph node size in locally advanced cervical cancer treated with concurrent chemoradiotherapy. Yeungnam Univ J Med. 2019 May;36(2):115-123. doi: 10.12701/yujm.2019.00143. Epub 2019 Feb 21. PMID 31620623
- [Background] Pedone Anchora L, Carbone V, Gallotta V, Fanfani F, Cosentino F, Turco LC, Fedele C, Bizzarri N, Scambia G, Ferrandina G. Should the Number of Metastatic Pelvic Lymph Nodes be Integrated into the 2018 Figo Staging Classification of Early Stage Cervical Cancer? Cancers (Basel). 2020 Jun 12;12(6):1552. doi: 10.3390/cancers12061552. PMID 32545508
- [Background] Zhou J, Wu SG, Sun JY, Liao XL, Li FY, Lin HX, Yang LC, He ZY. Incorporation of the number of positive lymph nodes leads to better prognostic discrimination of node-positive early stage cervical cancer. Oncotarget. 2017 Apr 18;8(16):26057-26065. doi: 10.18632/oncotarget.15220. PMID 28199962
- [Background] Wang SC, Lin LC, Kuo YT, Lin YW. Radiographic Number of Positive Pelvic Lymph Nodes as a Prognostic Factor in Cervical Cancer Treated With Definitive Concurrent Chemoradiotherapy or Intensity-Modulated Radiotherapy. Front Oncol. 2018 Nov 30;8:546. doi: 10.3389/fonc.2018.00546. eCollection 2018. PMID 30555798
- [Background] Tohyama A, Murakami M, Yoshino K. Strategies for the Treatment of Cervical Cancer with Bulky Pelvic Lymph Nodes: An Overview of the Current Evidence. J UOEH. 2020;42(4):317-325. doi: 10.7888/juoeh.42.317. PMID 33268608
- [Background] Marnitz S, Kohler C, Roth C, Fuller J, Hinkelbein W, Schneider A. Is there a benefit of pretreatment laparoscopic transperitoneal surgical staging in patients with advanced cervical cancer? Gynecol Oncol. 2005 Dec;99(3):536-44. doi: 10.1016/j.ygyno.2005.07.005. Epub 2005 Aug 29. PMID 16126259
- [Background] Yang J, Delara R, Magrina J, Magtibay P, Yi J, Langstraat C, Robertson M, Dinh T, Butler K. Comparing survival outcomes between surgical and radiographic lymph node assessment in locally advanced cervical cancer: A propensity score-matched analysis. Gynecol Oncol. 2020 Feb;156(2):320-327. doi: 10.1016/j.ygyno.2019.12.009. Epub 2019 Dec 14. PMID 31843274
- [Background] Lee M, Choi CH, Chun YK, Kim YH, Lee KB, Lee SW, Shim SH, Song YJ, Roh JW, Chang SJ, Lee JM. Surgical manual of the Korean Gynecologic Oncology Group: classification of hysterectomy and lymphadenectomy. J Gynecol Oncol. 2017 Jan;28(1):e5. doi: 10.3802/jgo.2017.28.e5. Epub 2016 Aug 19. PMID 27670259
- [Background] Shin W, Ham TY, Park YR, Lim MC, Won YJ. Comparing survival outcomes for cervical cancer based on the 2014 and 2018 International Federation of Gynecology and Obstetrics staging systems. Sci Rep. 2021 Mar 26;11(1):6988. doi: 10.1038/s41598-021-86283-2. PMID 33772044
- [Background] Lim MC, Bae J, Park JY, Lim S, Kang S, Seo SS, Kim JY, Rho JW, Park SY. Experiences of pretreatment laparoscopic surgical staging in patients with locally advanced cervical cancer: results of a prospective study. J Gynecol Oncol. 2008 Jun;19(2):123-8. doi: 10.3802/jgo.2008.19.2.123. Epub 2008 Jun 20. PMID 19471562
- [Background] Lorusso D, Xiang Y, Hasegawa K, Scambia G, Leiva M, Ramos-Elias P, Acevedo A, Cvek J, Randall L, Pereira de Santana Gomes AJ, Contreras Mejia F, Helpman L, Akilli H, Lee JY, Saevets V, Zagouri F, Gilbert L, Sehouli J, Tharavichitkul E, Lindemann K, Colombo N, Chang CL, Bednarikova M, Zhu H, Oaknin A, Christiaens M, Petru E, Usami T, Liu P, Yamada K, Toker S, Keefe SM, Pignata S, Duska LR; ENGOT-cx11/GOG-3047/KEYNOTE-A18 investigators. Pembrolizumab or placebo with chemoradiotherapy followed by pembrolizumab or placebo for newly diagnosed, high-risk, locally advanced cervical cancer (ENGOT-cx11/GOG-3047/KEYNOTE-A18): overall survival results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Oct 5;404(10460):1321-1332. doi: 10.1016/S0140-6736(24)01808-7. Epub 2024 Sep 14. PMID 39288779
- [Background] Manders DB, Sims TT, Bailey A, Hwang L, Richardson DL, Miller DS, Kehoe SM, Albuquerque KV, Lea JS. The Significance of Para-Aortic Nodal Size and the Role of Adjuvant Systemic Chemotherapy in Cervical Cancer: An Institutional Experience. Am J Clin Oncol. 2018 Dec;41(12):1225-1230. doi: 10.1097/COC.0000000000000458. PMID 29782361
- [Background] Kodama J, Seki N, Ojima Y, Nakamura K, Hongo A, Hiramatsu Y. Prognostic factors in node-positive patients with stage IB-IIB cervical cancer treated by radical hysterectomy and pelvic lymphadenectomy. Int J Gynaecol Obstet. 2006 May;93(2):130-5. doi: 10.1016/j.ijgo.2006.02.012. Epub 2006 Mar 6. PMID 16563395
- [Background] Park JW, Bae JW. Prognostic significance of positive lymph node number in early cervical cancer. Mol Clin Oncol. 2016 Jun;4(6):1052-1056. doi: 10.3892/mco.2016.837. Epub 2016 Mar 30. PMID 27284443
- [Background] Inoue T, Morita K. The prognostic significance of number of positive nodes in cervical carcinoma stages IB, IIA, and IIB. Cancer. 1990 May 1;65(9):1923-7. doi: 10.1002/1097-0142(19900501)65:93.0.co;2-m. PMID 2372764
- [Background] Sakuragi N, Satoh C, Takeda N, Hareyama H, Takeda M, Yamamoto R, Fujimoto T, Oikawa M, Fujino T, Fujimoto S. Incidence and distribution pattern of pelvic and paraaortic lymph node metastasis in patients with Stages IB, IIA, and IIB cervical carcinoma treated with radical hysterectomy. Cancer. 1999 Apr 1;85(7):1547-54. doi: 10.1002/(sici)1097-0142(19990401)85:73.0.co;2-2. PMID 10193945
- [Background] Kato T, Watari H, Takeda M, Hosaka M, Mitamura T, Kobayashi N, Sudo S, Kaneuchi M, Kudo M, Sakuragi N. Multivariate prognostic analysis of adenocarcinoma of the uterine cervix treated with radical hysterectomy and systematic lymphadenectomy. J Gynecol Oncol. 2013 Jul;24(3):222-8. doi: 10.3802/jgo.2013.24.3.222. Epub 2013 Jul 4. PMID 23875071
- [Background] Kim JH, Choi JH, Ki EY, Lee SJ, Yoon JH, Lee KH, Park TC, Park JS, Bae SN, Hur SY. Incidence and risk factors of lower-extremity lymphedema after radical surgery with or without adjuvant radiotherapy in patients with FIGO stage I to stage IIA cervical cancer. Int J Gynecol Cancer. 2012 May;22(4):686-91. doi: 10.1097/IGC.0b013e3182466950. PMID 22398707
- [Background] Lee J, Byun HK, Im SH, Son WJ, Roh YH, Kim YB. Risk factors for lower extremity lymphedema after surgery in cervical and endometrial cancer. J Gynecol Oncol. 2023 May;34(3):e28. doi: 10.3802/jgo.2023.34.e28. Epub 2022 Dec 19. PMID 36562134
- [Background] Carlson JW, Kauderer J, Hutson A, Carter J, Armer J, Lockwood S, Nolte S, Stewart BR, Wenzel L, Walker J, Fleury A, Bonebrake A, Soper J, Mathews C, Zivanovic O, Richards WE, Tan A, Alberts DS, Barakat RR. GOG 244-The lymphedema and gynecologic cancer (LEG) study: Incidence and risk factors in newly diagnosed patients. Gynecol Oncol. 2020 Feb;156(2):467-474. doi: 10.1016/j.ygyno.2019.10.009. Epub 2019 Dec 16. PMID 31837831
- [Background] Borcinova M, Ragosch V, Jarkovsky J, Bajsova S, Pilka R, Glickman A, Garrido-Mallach S, Raspagliesi F, Szatkowski W, Pakiz M, Snyman LC, Kocian R, Tamussino K, Kalist V, Michal M, Segovia MG, Poka R, Kipp B, Szewczyk G, Wydra D, Toth R, Vinnytska A, Fischerova D, Siegler K, Cibula D. Challenges in lower limb lymphoedema assessment based on limb volume change: Lessons learnt from the SENTIX prospective multicentre study. Gynecol Oncol. 2022 Jan;164(1):76-84. doi: 10.1016/j.ygyno.2021.10.089. Epub 2021 Nov 8. PMID 34763939
- [Background] Devoogdt N, Lemkens H, Geraerts I, Van Nuland I, Flour M, Coremans T, Christiaens MR, Van Kampen M. A new device to measure upper limb circumferences: validity and reliability. Int Angiol. 2010 Oct;29(5):401-7. PMID 20924341
- [Derived] Yun BS, Lee KB, Lee KH, Chang HK, Kim JY, Lim MC, Choi CH, Cho H, Kim DY, Kim YH, Choi JS, Lee CH, Kim JW, Kim SW, Kim YB, Cho CH, Hong DG, Song YJ, Jeon S, Kim MK, Jeong DH, Park H, Kim SM, Park SI, Song JY, Mukhopadhyay A, Thinh DHQ, Kampan NC, Lee GJ, Kim JH, Eom KY, Roh JW; Korean Gynecologic Oncology Group (KGOG) Investigators. Therapeutic effects of surgical debulking of metastatic lymph nodes in cervical cancer IIICr: a trial protocol for a phase III, multicenter, randomized controlled study (KGOG1047/DEBULK trial). J Gynecol Oncol. 2024 Sep;35(5):e57. doi: 10.3802/jgo.2024.35.e57. Epub 2024 Jan 22. PMID 38330380
- See also: L. Framework, Best practice for the management of lymphoedema, International consensus, MEP Ltd, London, 2006. — https://www.lympho.org/uploads/files/files/Best_practice.pdf